CLINICAL TRIAL: NCT06699225
Title: Investigation of Knowledge and Practices Regarding Pediatric Osteoporosis in Türkiye: A Cross-Sectional Study
Brief Title: Investigation of Knowledge and Practices Regarding Pediatric Osteoporosis in Türkiye
Acronym: PedOp
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, MD, Medical doctor, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: 2024/24-703
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis; Pediatric
Keywords: pediatric osteoporosis; knowlage assesment tool; pm&r; pediatry; orthopedics
MeSH Terms: conditions — Osteoporosis; Juvenile osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational- cross sectional study is to investigate the knowledge and practices of physicians in Physical Medicine and Rehabilitation (PM&R), Pediatrics, and Orthopedics regarding pediatric osteoporosis. The main question it aims to answer is:

What are the levels of knowledge and approaches of physicians in PM&R, Pediatrics, and Orthopedics regarding pediatric osteoporosis, and how can a psychometrically valid and reliable data collection tool be developed to measure these?

Participants, including PM&R, Pediatrics, and Orthopedics physicians, will complete an online questionnaire consisting of demographic and clinical practice questions, as well as items measuring their knowledge about pediatric osteoporosis. The study also includes a pilot test with a subset of participants to evaluate the clarity and reliability of the questionnaire.

DETAILED DESCRIPTION:
The aim of this study was to investigate the knowledge and approaches of physicians in Physical Medicine and Rehabilitation (PM&R), Pediatrics, and Orthopedics regarding pediatric osteoporosis. A secondary aim was to develop and evaluate the psychometric properties of a data collection tool designed to measure knowledge and practices related to pediatric osteoporosis.

The Pediatric Osteoporosis Knowledge and Practice Assessment Scale, used as the data collection tool, was developed based on evidence-based guidelines and the International Society for Clinical Densitometry Pediatric Position Statements. The scale consists of a preliminary section assessing demographic data and clinical practices, and a second section measuring knowledge levels. The questions were designed with "true" (1 point), "false," and "I don't know" (0 points) options, similar to the Osteoporosis Knowledge Questionnaire, which is intended for adults. The questions were categorized into general knowledge and diagnosis, risk factors, assessment, and treatment.

Content validity of the scale was ensured by a panel of experts in the field. The scale was distributed online via Google Forms and applied to 321 physicians. A pilot test was conducted with 10 PM&R physicians to evaluate its clarity. To assess reliability, the scale was administered twice to 30 physicians with a one-week interval.

ELIGIBILITY:
Inclusion Criteria:

* Physicians specializing in Physical Medicine and Rehabilitation (PM&R), Pediatrics, or Orthopedics
* Able to read and understand the language in which the questionnaire is provided,
* Internet access to complete the online survey distributed via Google Forms
* Willing to participate and provide informed consent
* Actively practicing in their respective specialty.
* Involved in the care of patients where knowledge about pediatric osteoporosis is relevant

Exclusion Criteria:

* Surveys with incomplete or inconsistent answers that do not meet the study's data quality standards
* Participants who have been involved in the development or validation of the Pediatric Osteoporosis Knowledge and Practice Assessment Scale

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of licensed physicians specializing in Physical Medicine and Rehabilitation (PM&R), Pediatrics, and Orthopedics who are actively practicing and involved in the care of patients where knowledge about pediatric osteoporosis is relevant.
  Participants are recruited online through professional networks, medical organizations, and personal invitations. The study is conducted using an online survey format to ensure accessibility and convenience for participants. The target population includes both early-career and experienced physicians to comprehensively assess the knowledge and practices across different levels of expertise.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Level of knowledge and practices of physicians in Physical Medicine and Rehabilitation (PM&R), Pediatrics, and Orthopedics regarding pediatric osteoporosis. | From October 2024 to November 2024
  This outcome will likely be measured by:
  The total score obtained from the Pediatric Osteoporosis Knowledge and Practice Assessment Scale, which evaluates knowledge in the domains of general information and diagnosis, risk factors, assessment, and treatment.

SECONDARY OUTCOMES:
Validation and reliability of the Pediatric Osteoporosis Knowledge and Practice Assessment Scale as a psychometric tool | From October 2024 to November 2024
  This will be assessed through:
  Reliability Testing:
  Test-retest reliability using the Intraclass Correlation Coefficient (ICC) from responses collected one week apart.
  Internal Consistency:
  Cronbach's alpha coefficient to determine the consistency of the items within the scale.
  Structural Validity:
  Factor analysis to confirm that the scale items align with predefined theoretical domains (e.g., general knowledge and diagnosis, risk factors, assessment, and treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Aslinur Keles Ercisli, Principal Investigator — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided